CLINICAL TRIAL: NCT00742924
Title: Feasibility and Dose Discovery Analysis of Zoledronic Acid With Concurrent Chemotherapy in the Treatment of Newly Diagnosed Metastatic Osteosarcoma
Brief Title: Zoledronic Acid and Combination Chemotherapy in Treating Patients With Newly Diagnosed Metastatic Osteosarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOST06P1; CDR0000612613 (Other: Clinical Trials.gov); COG-AOST06P1 (Other: Children's Oncology Group)
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-06

CONDITIONS: Sarcoma
Keywords: metastatic osteosarcoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma | interventions — Cisplatin; Dexrazoxane; Razoxane; Doxorubicin; Etoposide; etoposide phosphate; Ifosfamide; Leucovorin; Methotrexate; Zoledronic Acid; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Filgrastim; Granulocyte Colony-Stimulating Factor; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1- Chemotherapy and 1.2 mg/m2 Zoledronic Acid (Experimental): (Weeks 1-11) Patients receive dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; and G-CSF SC. (Week 12) Patients undergo therapeutic conventional surgery .
  (Weeks 13-25): Patients receive etoposide IV; ifosfamide IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; G-CSF SC. (Week 26) Patients may undergo surgical procedure.
  (Weeks 27-36): Patients receive dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; etoposide IV; ifosfamide IV; and filgrastim (G-CSF) SC.
  See Detailed Description.
  Interventions: Drug: cisplatin; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: leucovorin calcium; Drug: methotrexate; Drug: zoledronic acid; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery; Biological: filgrastim; Drug: Mesna
- Arm 2 - Chemotherapy and 2.3 mg/m2 Zoledronic Acid (Experimental): (Weeks 1-11) Patients receive dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; and G-CSF SC. (Week 12) Patients undergo therapeutic conventional surgery.
  (Weeks 13-25): Patients receive etoposide IV; ifosfamide IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; G-CSF SC. (Week 26) Patients may undergo surgical procedure.
  (Weeks 27-36): Patients receive dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; etoposide IV; ifosfamide IV; and filgrastim (G-CSF) SC.
  See Detailed Description.
  Interventions: Drug: cisplatin; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: leucovorin calcium; Drug: methotrexate; Drug: zoledronic acid; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery; Biological: filgrastim; Drug: Mesna
- Arm 3 - Chemotherapy and 3.5 mg/m2 Zoledronic Acid (Experimental): (Weeks 1-11) Patients receive dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; and G-CSF SC. (Week 12) Patients undergo therapeutic conventional surgery.
  (Weeks 13-25): Patients receive etoposide IV; ifosfamide IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; G-CSF SC. (Week 26) Patients may undergo surgical procedure.
  (Weeks 27-36): Patients receive dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; etoposide IV; ifosfamide IV; and filgrastim (G-CSF) SC.
  See Detailed Description.
  Interventions: Drug: cisplatin; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: leucovorin calcium; Drug: methotrexate; Drug: zoledronic acid; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery; Biological: filgrastim; Drug: Mesna
- Chemotherapy and 2.3 mg/m2 Zoledronic Acid after MTD (Experimental): (Weeks 1-11) Patients receive dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; and G-CSF SC. (Week 12) Patients undergo therapeutic conventional surgery.
  (Weeks 13-25): Patients receive etoposide IV; ifosfamide IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; G-CSF SC. (Week 26) Patients may undergo surgical procedure.
  (Weeks 27-36): Patients receive dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; etoposide IV; ifosfamide IV; and filgrastim (G-CSF) SC.
  See Detailed Description.
  Interventions: Drug: cisplatin; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: leucovorin calcium; Drug: methotrexate; Drug: zoledronic acid; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery; Biological: filgrastim; Drug: Mesna

INTERVENTIONS:
Drug: cisplatin — Given IV
  Other Names: Cis-diamminedichloroplatinum II; CDDP; cis-DDP; Platinol-AQ; NSC #119875
Drug: dexrazoxane hydrochloride — Given IV
  Other Names: ICRF-187; ADR-529; ZINECARD; NSC #169780
Drug: doxorubicin hydrochloride — Given IV
  Other Names: Adriamycin; NSC #123127
Drug: etoposide — Given IV
  Other Names: VePesid; Etopophos; VP-16; NSC #141540
Drug: ifosfamide — Given IV
  Other Names: Isophosphamide; Iphosphamide; Z4942; Ifex; NSC #109724
Drug: leucovorin calcium — Given IV or orally
  Other Names: LCV; Wellcovorin; citrovorum factor; folinic acid; NSC #003590
Drug: methotrexate — Given IV
  Other Names: MTX; amethopterin; Trexall; NSC #000740
Drug: zoledronic acid — Given IV
  Other Names: 1-Hydroxy-2-imidazol-1-ylethylidene - diphosphonic acid; zoledronate; Zometa; Aclasta; NSC# 721517
Procedure: adjuvant therapy
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery — Surgery of the primary tumor is scheduled for 12 weeks after the commencement of chemotherapy.
Biological: filgrastim — Given SC
  Other Names: Granulocyte Colony-Stimulating Factor; r-metHuG-CSF; G-CSF; Neupogen; NSC #614629
Drug: Mesna — Given IV
  Other Names: sodium 2-mercaptoethane sulfonate; UCB 3983; Mesnex; NSC #113891

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This clinical trial is studying the side effects and best dose of zoledronic acid when given together with combination chemotherapy in treating patients with newly diagnosed metastatic osteosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary:

* To assess the feasibility and safety of zoledronic acid when administered in combination with standard chemotherapy in patients with newly diagnosed metastatic osteosarcoma.
* To determine the maximum tolerated dose of zoledronic acid when administered in combination with standard chemotherapy in these patients.

Secondary:

- To compare the histologic response and event-free survival of patients treated with this regimen versus patients treated on INT-0133 or CCG-7943.

OUTLINE: This is a multicenter, dose-escalation study of zoledronic acid.

* Induction therapy (weeks 1-11): Patients receive dexrazoxane hydrochloride IV slowly over 5-15 minutes, doxorubicin hydrochloride IV over 15 minutes, and cisplatin IV over 1 hour on days 1 and 2 of weeks 1 and 6; zoledronic acid IV at the assigned dose level over 30 minutes on day 4 of weeks 1 and 6; high-dose methotrexate IV over 4 hours on day 1 of weeks 4, 5, 9, and 10; leucovorin calcium IV or orally every 6 hours starting on day 2 and continuing until clearance of methotrexate of weeks 4, 5, 9, and 10; and filgrastim (G-CSF) subcutaneously (SC) once daily beginning on day 3 of weeks 1 and 6 and continuing until blood counts recover.
* Surgery (week 12): Patients undergo definitive surgery (limb-salvage surgery or amputation) of the primary tumor in week 12.
* Maintenance therapy course 1 (weeks 13-25): Patients receive etoposide IV over 1 hour and ifosfamide IV over 4 hours on days 1-5 of weeks 13 and 21; zoledronic acid IV over 30 minutes on day 4 of week 17 and on day 7 of weeks 13 and 21; high-dose methotrexate IV over 4 hours on day 1 of weeks 16, 20, and 24; leucovorin calcium IV or orally every 6 hours starting on day 2 and continuing until clearance of methotrexate of weeks 16, 20, and 24; dexrazoxane hydrochloride IV slowly over 5-15 minutes, doxorubicin hydrochloride IV over 15 minutes, and cisplatin IV over 1 hour on days 1 and 2 of week 17; and G-CSF SC once daily beginning on day 6 of weeks 13, 17, and 21 and continuing until blood counts recover.
* Surgery (week 26): Patients may undergo surgical resection of primary metastases in week 26.
* Maintenance therapy course 2 (weeks 27-36): Patients receive dexrazoxane hydrochloride IV slowly over 5-15 minutes and doxorubicin hydrochloride IV over 15 minutes on days 1 and 2 of weeks 27 and 31; cisplatin IV over 1 hour on days 1 and 2 of week 27; zoledronic acid IV over 30 minutes on day 4 of week 27 and on day 7 of weeks 31 and 36; high-dose methotrexate IV over 4 hours on day 1 of weeks 30, 34, and 35; leucovorin calcium IV or orally every 6 hours starting on day 2 and continuing until clearance of methotrexate of weeks 30, 34, and 35; etoposide IV over 1 hour on days 1-5 of week 36; ifosfamide (1.8 gm/m2 ) IV over 1 hour on days 1-5 of week 31;ifosfamide (2.8 gm/m2)IV over 4 hours on days 1-5 of week 36; and G-CSF SC once daily beginning on day 3 of weeks 27, 31, and 36 and continuing until blood counts recover.

Mensa is a supportive care medicine used to prevent hemorrhagic cystitis caused by ifosfamide. It is always given when ifosfamide is given. It was used in all arms.

After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven high-grade osteosarcoma within the past 6 weeks

  * Newly diagnosed disease
  * Metastatic disease
* Resectable disease OR expected to become resectable after initial chemotherapy
* Disease has arisen outside of areas of Paget's disease

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 50-100% (for patients > 16 years of age) OR Lansky PS 50-100% (for patients ≤ 16 years of age)
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR maximum serum creatinine based on age/gender as follows:

  * 0.4 mg/dL (for patients 1 to 5 months of age)
  * 0.5 mg/dL (for patients 6 to 11 months of age)
  * 0.6 mg/dL (for patients 1 year of age)
  * 0.8 mg/dL (for patients 2 to 5 years of age)
  * 1 mg/dL (for patients 6 to 9 years of age)
  * 1.2 mg/dL (for patients 10 to 12 years of age)
  * 1.5 mg/dL (males) or 1.4 mg/dL (females) (for patients 13 to 15 years of age)
  * 1.7 mg/dL (males) or 1.4 mg/dL (females) (for patients ≥ 16 years of age)
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN) for age
* AST or ALT < 2.5 times ULN for age
* Shortening fraction ≥ 28% by echocardiogram OR ejection fraction ≥ 50% by radionuclide angiogram
* ANC ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³ (transfusion independent)
* Hemoglobin ≥ 10 g/dL (RBC transfusion allowed)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use contraception
* No known HIV infection
* No history of pericarditis, myocarditis, symptomatic arrhythmia, or conduction disturbances

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy
* No other concurrent anticancer chemotherapy
* No concurrent immunomodulating agents
* Steroids for anti-emetic allowed

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2008-08; Primary Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Goldsby, MD, Study Chair — University of California, San Francisco
Locations (88):
- United States (77):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Keyser Family Cancer Center at Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Maine Children's Cancer Program at Barbara Bush Children's Hospital, Scarborough, Maine
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's - Dayton, Dayton, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - T.C. Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (9):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
- San Jorge Children's Hospital, Santurce, Puerto Rico

REFERENCES:
- [Derived] Goldsby RE, Fan TM, Villaluna D, Wagner LM, Isakoff MS, Meyer J, Randall RL, Lee S, Kim G, Bernstein M, Gorlick R, Krailo M, Marina N. Feasibility and dose discovery analysis of zoledronic acid with concurrent chemotherapy in the treatment of newly diagnosed metastatic osteosarcoma: a report from the Children's Oncology Group. Eur J Cancer. 2013 Jul;49(10):2384-91. doi: 10.1016/j.ejca.2013.03.018. Epub 2013 May 7. PMID 23664013

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1- Chemotherapy and 1.2 mg/m2 Zoledronic Acid: (Weeks 1-11) Patients receive dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; and G-CSF SC. (Week 12) Patients undergo therapeutic conventional surgery .
  (Weeks 13-25): Patients receive etoposide IV; ifosfamide IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; G-CSF SC. (Week 26) Patients may undergo surgical procedure.
  (Weeks 27-36): Patients receive dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; etoposide IV; ifosfamide IV; and filgrastim (G-CSF) SC.
  See Detailed Description.
  cisplatin: Given IV
  dexrazoxane hydrochloride: Given IV
  doxorubicin hydrochloride: Given IV
  etoposide: Given IV
  ifosfamide: Given IV
  leucovorin calcium: Given IV or orally
- Arm 2 - Chemotherapy and 2.3 mg/m2 Zoledronic Acid; Arm 3 - Chemotherapy and 3.5 mg/m2 Zoledronic Acid: (Weeks 1-11) Patients receive dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; and G-CSF SC. (Week 12) Patients undergo therapeutic conventional surgery.
  (Weeks 13-25): Patients receive etoposide IV; ifosfamide IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; G-CSF SC. (Week 26) Patients may undergo surgical procedure.
  (Weeks 27-36): Patients receive dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; etoposide IV; ifosfamide IV; and filgrastim (G-CSF) SC.
  See Detailed Description.
  cisplatin: Given IV
  dexrazoxane hydrochloride: Given IV
  doxorubicin hydrochloride: Given IV
  etoposide: Given IV
  ifosfamide: Given IV
  leucovorin calcium: Given IV or orally
- Chemotherapy and 2.3 mg/m2 Zoledronic Acid After MTD: (Weeks 1-11) Patients receive dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; and G-CSF SC. (Week 12) Patients undergo therapeutic conventional surgery.(Weeks 13-25): Patients receive etoposide IV; ifosfamide IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; G-CSF SC. (Week 26) Patients may undergo surgical procedure.(Weeks 27-36): Patients receive dexrazoxane hydrochloride IV; doxorubicin hydrochloride IV; cisplatin IV; zoledronic acid IV; high-dose methotrexate IV; leucovorin calcium IV or orally; etoposide IV; ifosfamide IV; and filgrastim (G-CSF) SC.See Detailed Description.
  cisplatin: Given IV
  dexrazoxane hydrochloride: Given IV
  doxorubicin hydrochloride: Given IV
  etoposide: Given IV
  ifosfamide: Given IV
  leucovorin calcium: Given IV or orally
Period: Overall Study
Arm/Group | Arm 1- Chemotherapy and 1.2 mg/m2 Zoledronic Acid | Arm 2 - Chemotherapy and 2.3 mg/m2 Zoledronic Acid | Arm 3 - Chemotherapy and 3.5 mg/m2 Zoledronic Acid | Chemotherapy and 2.3 mg/m2 Zoledronic Acid After MTD
Started | 6 | 6 | 6 | 6
Completed | 1 | 4 | 2 | 0
Not Completed | 5 | 2 | 4 | 6
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 5 | 1 | 2 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1- Chemotherapy and 1.2 mg/m2 Zoledronic Acid | Arm 2 - Chemotherapy and 2.3 mg/m2 Zoledronic Acid | Arm 3 - Chemotherapy and 3.5 mg/m2 Zoledronic Acid | Chemotherapy and 2.3 mg/m2 Zoledronic Acid After MTD | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Median (Full Range); unit: years] | 11.5 [8 to 20] | 15.5 [9 to 21] | 14 [10 to 19] | 14.5 [7 to 22] | 13.5 [7 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 2 | 5 | 16
  Male | 1 | 2 | 4 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 3 | 1 | 7
  White | 4 | 4 | 2 | 3 | 13
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 6 | 5 | 5 | 4 | 20
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 5 | 6 | 20
  Canada | 2 | 1 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Limiting Toxicity
Description: The occurrence of Limiting Toxicity defined as Any CTC AE version 4 Grade 3 and 4 non-hematologic toxicity thought to be possibly, probably or definitely related to zoledronic acid with the specific exclusion of:
  * Grade 3 nausea and vomiting controlled with adequate antiemetic prophylaxis.
  * Grade 3 transaminase (AST/ALT) that occurs during the evaluation period but resolves to ≤ Grade 2, before the planned dose of therapy after definitive surgery.
  * Grade 3 fever or infection.
  * Grade 3 or 4 hypocalcemia (see Section 5.1.1)
  * Grade 3 mucositis.
  * Grade 3 fatigue that returns to ≤ Grade 2, before the planned dose of therapy after definitive surgery.
  * Grade 3 joint range of motion, decreased or joint effusion that is related to the primary tumor.
Time Frame: Enrollment through the first 12 weeks of therapy.
Population: Patients found not to meet the eligibility requirements are by group policy not followed for adverse events or outcome
Measure: Number; unit: participants
Arm/Group | Arm 1- Chemotherapy and 1.2 mg/m2 Zoledronic Acid | Arm 2 - Chemotherapy and 2.3 mg/m2 Zoledronic Acid | Arm 3 - Chemotherapy and 3.5 mg/m2 Zoledronic Acid | Chemotherapy and 2.3 mg/m2 Zoledronic Acid After MTD
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants | 1 | 1 | 3 | 2

2. Secondary Outcome: Histologic Response as Assessed in the Primary Tumor and in Resected Metastases
Description: Histologic response as graded according to the system of Huvos across all specimens resected at the time of local control in the primary tumor and in resected metastases.
  The best response, as quantified by maximum necrosis grading according to the system of Huvos across all specimens resected at the time of local control, will be used to quantify the effect of Induction chemotherapy.
Time Frame: At definitive surgery planned for 12 weeks after the start of protocol therapy.
Reporting Status: Not Posted

3. Secondary Outcome: Event-free Survival
Description: The EFS and survival functions will be estimated by the Kaplan-Meier methodology.
Time Frame: Time from study enrollment to disease recurrence, death without disease progression, diagnosis of a second malignant neoplasm, assessed up to 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Secondary Limiting Toxicity
Description: Secondary limiting toxicity defined as Any CTC AE version 4 Grade 3 and 4 non-hematologic toxicity thought to be possibly, probably or definitely related to zoledronic acid with the specific exclusion of:
  * Grade 3 nausea and vomiting controlled with adequate antiemetic prophylaxis.
  * Grade 3 transaminase (AST/ALT) that occurs during the evaluation period but resolves to ≤ Grade 2, before the planned dose of therapy after definitive surgery.
  * Grade 3 fever or infection.
  * Grade 3 or 4 hypocalcemia (see Section 5.1.1)
  * Grade 3 mucositis.
  * Grade 3 fatigue that returns to ≤ Grade 2, before the planned dose of therapy after definitive surgery.
  * Grade 3 joint range of motion, decreased or joint effusion that is related to the primary tumor.
  CTC AE version 4 hematologic toxicity will be based on time to blood count recovery to an ANC ≥ 1000/µL and platelet count ≥ 100,000/µL that delays definitive surgery by more than 2 weeks.
Time Frame: After week 13 to the end of protocol therapy
Reporting Status: Not Posted

5. Secondary Outcome: Prognostic Value of Bone Resorption Markers
Description: Blood will be collected for quantification of c-telopeptide and urine will be collected for quantification of n-telopeptide.
Time Frame: At baseline and at weeks 13 and 36
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Arm 1- Chemotherapy and 1.2 mg/m2 Zoledronic Acid | Arm 2 - Chemotherapy and 2.3 mg/m2 Zoledronic Acid | Arm 3 - Chemotherapy and 3.5 mg/m2 Zoledronic Acid | Chemotherapy and 2.3 mg/m2 Zoledronic Acid After MTD
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1- Chemotherapy and 1.2 mg/m2 Zoledronic Acid (N=6) | Arm 2 - Chemotherapy and 2.3 mg/m2 Zoledronic Acid (N=6) | Arm 3 - Chemotherapy and 3.5 mg/m2 Zoledronic Acid (N=6) | Chemotherapy and 2.3 mg/m2 Zoledronic Acid After MTD (N=6)
Alanine aminotransferase increased (Investigations) | 3 | 4 | 2 | 1
Anemia (Blood and lymphatic system disorders) | 3 | 4 | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Edema limbs (General disorders) | 1 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 2 | 6 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 3 | 3 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 2 | 2 | 2 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 2 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 3 | 5 | 4 | 3
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Platelet count decreased (Investigations) | 3 | 4 | 2 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
White blood cell decreased (Investigations) | 4 | 5 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No